CLINICAL TRIAL: NCT00167544
Title: A Randomized Trial of Hydrocortisone in Very Preterm Infants at High Risk for Neurologic and Pulmonary Impairments
Brief Title: Randomized Trial of Hydrocortisone in Very Preterm High-Risk Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Nehal Parikh, Associate Professor of Pediatrics, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: K23NS048152 (NIH); K23NS048152 (NIH); HSC-MS-05-0218
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-07

CONDITIONS: Bronchopulmonary Dysplasia; Encephalomalacia; Premature Birth
Keywords: Bronchopulmonary Dysplasia; Encephalomalacia; Brain injury; Neurosensory impairment; Corticosteroids; Anti-Inflammatory Agents; Extremely Low Birth Weight (ELBW) infants; Premature Birth; Magnetic Resonance Imaging
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Encephalomalacia; Premature Birth; Brain Injuries | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 1. Tapering dose of hydrocortisone every 12 h over 7 day period
  Interventions: Drug: Hydrocortisone
- 2 (Placebo Comparator): 2. Identical-appearing saline placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrocortisone — Hydrocortisone 3 mg/kg/d divided q 12h IV/PO tapered over 7 days
  Arms: 1
Drug: Placebo — Saline
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether treatment of very preterm infants at high-risk for lung and brain injury with low dose hydrocortisone results in improved pulmonary and neurologic outcomes.

DETAILED DESCRIPTION:
Hypothesis: Among extremely low birth weight infants (ELBW; BW ≤ 1000 g) at high risk for bronchopulmonary dysplasia (BPD) and neurologic impairments, those infants randomized to seven days of hydrocortisone will demonstrate increased total cerebral tissue volumes as compared to infants randomized to placebo.

Specific Aims: 1) To perform a pilot blinded randomized controlled trial of a 7-day regimen of low dose hydrocortisone in ELBW infants at high risk for BPD and neurosensory impairments and assess its effect on cerebral tissue volumes. 2) Evaluate and report 2 year neurodevelopmental outcomes.

Background and Significance: Bronchopulmonary dysplasia is a disease of arrested lung development and lung inflammation. It is primarily seen in ELBW infants. Neurological delay, including cerebral palsy and mental retardation, affect up to 40%-50% of surviving ELBW infants. BPD is an important risk factor for such neurological delay. Postnatal administration of corticosteroids to ventilated preterm neonates results in a reduced risk of developing BPD. Postnatal corticosteroids however have shown harmful effects on the brain and can lead to increased rates of cerebral palsy and learning problems. This effect has primarily been seen with dexamethasone when high doses were given in the first week of life. Beyond the first week of life, there is insufficient information on the effects of steroids on the brain. Steroids other than dexamethasone, in much lower doses have been shown to improve short term lung function with minimal short-term side effects. A review study of all steroid trials for BPD shows that when given to a high risk group of infants (> 50% risk of BPD) steroids protect the brain and reduce rates of cerebral palsy. The American and Canadian Pediatric societies and respected researchers have commented on the urgent need for more trials of other corticosteroids at lower doses started after the first week of life to evaluate their short and long-term pulmonary and neurological benefits and risks.

Research Design and Methods:

1. Inclusion & Exclusion Criteria: See below.
2. Procedures: Consented eligible patients will be randomly assigned to receive hydrocortisone in a tapering schedule over 7 days or placebo (comparison group). Study drug will be given every 12 hours IV with only study pharmacist aware of assignment. The patient's anatomic brain MRI (routinely done on all ELBW infants at 38 weeks post-menstrual age) will be further processed by the masked study investigators to derive total and regional brain volumes. Administration of indomethacin or dexamethasone to enrolled infants will be closely monitored and regulated throughout the trial period. Indomethacin use during study period is contraindicated. Dexamethasone (or other steroid) use will be restricted to ELBW infants on high ventilator settings (RIS > 10) after 28 days of life. All other procedures will be per routine care. Blinded developmental follow-up at two years, already currently performed for all ELBW infants at MHCH, will be analyzed and reported for all study infants.

ELIGIBILITY:
Inclusion Criteria:

* Patient in the Memorial Hermann Children's Hospital (MHCH) neonatal intensive care unit with a birth weight ≤ 1000 grams.
* Ventilator-dependent between 10 and 21 days of age.
* Respiratory index score (RIS: mean airway pressure x fraction of inspired oxygen) of ≥ 2.0 that is increasing or stable for the previous 24 hours or a RIS ≥ 3.0 if improvement noted in the past 24 hours.

Exclusion Criteria:

* Prior postnatal steroid treatment.
* Evidence of sepsis or necrotizing enterocolitis.
* Known major congenital anomalies of the cardiopulmonary or central nervous system.
* Infants being treated with indomethacin or those likely to require treatment in the next 7 days as judged by the treating physician.
* Inability or unwillingness of parent or legal guardian/representative to give written informed consent.
* Gestational age < 23 weeks.

Ages: 1 Week to 3 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2005-11; Primary Completion 2009-01 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nehal A. Parikh, D.O., M.S., Principal Investigator — The Research Institute at Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Parikh NA, Lasky RE, Kennedy KA, Moya FR, Hochhauser L, Romo S, Tyson JE. Postnatal dexamethasone therapy and cerebral tissue volumes in extremely low birth weight infants. Pediatrics. 2007 Feb;119(2):265-72. doi: 10.1542/peds.2006-1354. PMID 17272615
- [Background] Yu X, Zhang Y, Lasky RE, Datta S, Parikh NA, Narayana PA. Comprehensive brain MRI segmentation in high risk preterm newborns. PLoS One. 2010 Nov 8;5(11):e13874. doi: 10.1371/journal.pone.0013874. PMID 21079730
- [Result] Parikh NA, Kennedy KA, Lasky RE, McDavid GE, Tyson JE. Pilot randomized trial of hydrocortisone in ventilator-dependent extremely preterm infants: effects on regional brain volumes. J Pediatr. 2013 Apr;162(4):685-690.e1. doi: 10.1016/j.jpeds.2012.09.054. Epub 2012 Nov 8. PMID 23140612
- [Derived] Parikh NA, Kennedy KA, Lasky RE, Tyson JE. Neurodevelopmental Outcomes of Extremely Preterm Infants Randomized to Stress Dose Hydrocortisone. PLoS One. 2015 Sep 16;10(9):e0137051. doi: 10.1371/journal.pone.0137051. eCollection 2015. PMID 26376074
- See also: Patient information page - Bronchopulmonary Dysplasia — http://www.nhlbi.nih.gov/health/dci/Diseases/Bpd/Bpd_WhatIs.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All extremely low birth weight infants (ELBW; birth weight <=1000g) that were mechanically ventilated between day of life 10 to 21 were screened for eligibility in the neonatal intensive care unit at Children's Memorial Hermann Hospital during the period of October 11, 2005 and September 8, 2008.
Pre-assignment Details: Parent/guardian was approached if infant's respiratory index score (mean airway pressure x FiO2) was ≥ 2.0 and stable or increasing or if the respiratory index score was ≥ 3.0 when improvement was noted in the previous 24 hour period.
Groups:
- Hydrocortisone Arm: Subjects randomized by the investigational drug pharmacist to hydrocortisone arm received a 7 day course of intravenous (IV) hydrocortisone sodium succinate (Solu-Cortef) every 12 hours (3 mg/kg per day for first 4 days, 2 mg/kg per day for 2 days and 1 mg/kg per day for 1 day; total of 17 mg/kg over 7 days). The IV route was preferred.
- Placebo Arm: Subjects randomized by the investigational drug pharmacist to the placebo arm received an equivalent volume of identical appearing 0.9% sterile saline placebo. The IV route was preferred.
Period: Overall Study
Arm/Group | Hydrocortisone Arm | Placebo Arm
Started | 31 | 33
Completed | 30 | 33
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrocortisone Arm | Placebo Arm | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 33 | 64
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Median (Inter-Quartile Range); unit: weeks] — Gestational age
  weeks | 25 (3) [24 to 26] | 25 (3) [24 to 27] | 25 (3) [24 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 14 | 20 | 34
Region of Enrollment [Number; unit: participants]
  United States | 31 | 33 | 64

OUTCOME MEASURES:

1. Primary Outcome: Total Cerebral Volume as Measured by Volumetric Brain MRI
Description: Total cerebral volume included all brain gray matter and white matter, including cerebellum.
Time Frame: 38 weeks postmenstrual age (PMA)
Population: Eight infants died in each group prior to term MRI precluding a determination of brain volumes. Additionally, four infants had poor quality MRI scans that could not be analyzed for brain volumes.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Hydrocortisone Arm | Placebo Arm
Number analyzed (Participants) | 23 | 21
cm^3 | 272.01 (40.30) | 277.82 (59.05)

2. Secondary Outcome: Regional Brain Volumes
Description: Cerebral white matter volume
Time Frame: 38-weeks postmenstrual age
Population: In addition to the reasons cited for the primary outcome, one infant in the hydrocortisone group and two in the placebo group had artifacts on brain MRI precluding cerebral white matter segmentation and volume determination.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Hydrocortisone Arm | Placebo Arm
Number analyzed (Participants) | 22 | 19
cm^3 | 122.45 (18.73) | 118.62 (17.51)
Statistical Analysis 1: Comparison: Hydrocortisone Arm vs Placebo Arm; The primary analysis of total brain tissue volume was performed using multiple linear regression controlling for postmenstrual age at MRI scan to adjust for differences in timing at MRI. The distributions of potentially important confounding variables at baseline were compared in the two groups using parametric and non-parametric tests as appropriate. All analyses were performed using STATA 11.0. Please see PubMed: 23140612; Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Final Values) = 5.40, 95% CI 2-sided [-19.49 to 30.29]

3. Secondary Outcome: Duration of Positive Pressure Support (Mechanical Ventilation or Continuous Positive Airway Pressure)
Time Frame: Up to 36 weeks PMA
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Hydrocortisone Arm | Placebo Arm
Number analyzed (Participants) | 31 | 33
days | 68.7 [63.4 to 74.0] | 65.9 [59.7 to 72.0]

4. Secondary Outcome: Duration of Oxygen Requirement
Time Frame: Up to 36 weeks PMA
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Hydrocortisone Arm | Placebo Arm
Number analyzed (Participants) | 31 | 33
days | 72.7 [68.0 to 77.4] | 72.0 [66.9 to 77.1]

5. Secondary Outcome: Survival Without Severe Bronchopulmonary Dysplasia (BPD)
Description: Using the NIH Consensus definition (Jobe A, 2001)
Time Frame: 36 weeks postmenstrual age
Measure: Number; unit: participants
Arm/Group | Hydrocortisone Arm | Placebo Arm
Number analyzed (Participants) | 31 | 33
participants | 3 | 5

ADVERSE EVENTS:
Arm/Group | Hydrocortisone Arm | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 8/31 | 8/33
Other Adverse Events (participants affected / at risk) | 2/31 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocortisone Arm (N=31) | Placebo Arm (N=33)
Death before NICU discharge (Cardiac disorders) | 8 (8) | 8 (8)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocortisone Arm (N=31) | Placebo Arm (N=33)
Spontaneous intestinal perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No